CLINICAL TRIAL: NCT05098990
Title: A Prospective, Randomized, Multicenter Real-world Study of Jinfukang Oral Liquid Combined With Chemotherapy in Treatment for Patients With Driver Gene-negative Advanced Non-small Cell Lung Cancer
Brief Title: Jinfukang Oral Liquid Combined With Chemotherapy for Treating Driver Gene-negative Advanced NSCLC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Resources Sanjiu Medical & Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICM-JFK-CR01
Record Dates: First submitted 2021-09-21; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jinfukang oral liquid+Platinum-based doublet chemotherapy (Experimental): The usage cycle of Jinfukang oral liquid will be consistent with platinum-based doublet chemotherapy. Jinfukang oral liquid will be taken at day 5 after chemotherapy, and will be taken continuously 3 times per day and 30 mL per time at least 4 cycles. The usage of platinum-based doublet chemotherapy will be performed following the details described at the "Primary Lung Cancer Diagnosis and Treatment Guidelines" and "Chinese Society of Clinical Oncology (CSCO) Guidelines for the Diagnosis and Treatment of Non-small Cell Lung Cancer".
  Interventions: Drug: Jinfukang oral liquid
- Platinum-based doublet chemotherapy (Active Comparator): The usage of platinum-based doublet chemotherapy will be performed following the details described at the "Primary Lung Cancer Diagnosis and Treatment Guidelines" and "Chinese Society of Clinical Oncology (CSCO) Guidelines for the Diagnosis and Treatment of Non-small Cell Lung Cancer".
  Interventions: Drug: Platinum-based doublet chemotherapy

INTERVENTIONS:
Drug: Jinfukang oral liquid — Jinfukang koufuye is a Chinese herbal prescription, which is used in treatment for patients with NSCLC in clinical practice. It has been proved to be capable of preventing the occurrence of metastasis, stabilizing tumor lesions, improving the response rates when combined with chemotherapy, and prolonging the survival period of lung cancer patients.
  Other Names: Jinfukang koufuye
  Arms: Jinfukang oral liquid+Platinum-based doublet chemotherapy
Drug: Platinum-based doublet chemotherapy — Platinum-based doublet chemotherapy as first line therapy has been shown to be efficacious against non-small cell lung cancer.
  Other Names: Chemotherapy
  Arms: Platinum-based doublet chemotherapy

SUMMARY:
This is a prospective, randomized, multicenter real-world study, which aims to investigate the efficacy and safety of Jinfukang oral liquid combined with chemotherapy as first-line treatment regimen for patients with driver-negative advanced NSCLC. 328 patients with unresectable stage IIIB-IV NSCLC and Qi-Yin deficiency will be divided into experimental (n=164) and control groups (n=164) according to the stratified blocked randomization.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age;
2. Patients with stage ⅢB-IV NSCLC are diagnosed by histopathology and cytology;
3. Patients' tumor tissues are unresectable as assessed by the investigator;
4. Have measurable disease based on RECIST 1.1;
5. Driver gene (EGFR/ALK/ROS1) is negative;
6. Patients who are receiving first-line platinum-doublet chemotherapy with remaining no fewer than 4 therapeutic cycles;
7. Patients in chemotherapy who combined with other systemic therapy (including but not limited to immune checkpoint inhibitors and anti-vascular targeted drugs) are not suitable, but with radiotherapy can be permitted;
8. During chemotherapy cycles, patients who take prior treatment with anticancer Chinese medicine less than 4 weeks can be enrolled after stopping medication. If administration time is longer than 4 weeks, at least 4 weeks washout period should be performed;
9. Patients are diagnosed with Qi-yin deficiency by the Syndrome Differentiation of Traditional Chinese Medicine;
10. The expected survival time ≥3 months;
11. The subjects volunteer to sign the informed consent.

Exclusion Criteria:

1. Allergy or hypersensitivity to ingredients of the study treatment formulation;
2. Pregnant or lactating women;
3. Patients with multiple brain metastases, multiple bone metastases and liver metastases, which have great influence on survival times；
4. Patients are enrolling in other therapeutic trials;
5. The investigator does not consider the participant to be eligible for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2021-10-25 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 18 months
  Time from the start of treatment to first progression disease or death, whichever is earlier, according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 18 months
  Time from randomization to death from any cause, according to RECIST 1.1 criteria.
Objective Response Rate (ORR) | Up to 18 months
  ORR is defined as the percentage of subjects with confirmed best overall response of complete response (CR) or partial response (PR), according to RECIST 1.1 criteria.
Disease Control Rate (DCR) | Up to 18 months
  Disease control rate is defined as the proportion of patients with complete response (CR) or partial response (PR) or subjects with stable disease (SD), according to RECIST 1.1 criteria.
Quality of Life as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) | Up to 18 months
  30 quality of life questions for the participant to answer. The first 28 questions have answers that range from 1 (Not at All) to 4 (Very Much), and the final 2 questions answers range from 1 (Very Poor) to 7 (Excellent).
Quality of Life as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire LC-13 (EORTC QLQ-LC13) | Up to 18 months
  13 quality of life questions for the participant to answer. The answers range from 1 (Not at All) to 4 (Very Much).
Incidence and Severity of Adverse Events (AE) | Up to 18 months
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Incidence and Severity of Serious Adverse Event (SAE) | Up to 18 months
  SAE refers to events that require hospitalization, prolong hospitalization, disability, impact on work ability, life-threatening or death, and congenital malformations that occur during clinical trials.
Incidence and severity of Adverse Drug Reactions (ADR)，Serious Adverse Drug Reactions (SADR) or Suspected Unexpected Serious Adverse Drug Reactions (SUSAR) | Up to 18 months
  ADR: All noxious and unintended responses to a medicinal product related to any dose. SUSAR: all suspected adverse.
Change from baseline of peripheral immune cell counts | Up to 18 months
  Surface expression of CD3, CD4 and CD8 is assessed as a marker of absolute T lymphocyte, T helper cell and cytotoxic T lymphocyte, respectively.

OTHER OUTCOMES:
Circulating tumor DNA (ctDNA) level measurement | Up to 18 months
  Blood sample will be collected for ctDNA testing.